CLINICAL TRIAL: NCT02329977
Title: Rate of Duodenal-biliary Reflux Increases in Patients With Recurrent Common Bile Duct Stones: Direct Evidence From Barium Meal Examination
Brief Title: Rate of Duodenal-biliary Reflux Increases in Patients With Recurrent Common Bile Duct Stones
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20130508-2
Record Dates: First submitted 2014-12-20; First posted 2015-01-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Common Bile Duct Gall Stones; Common Bile Duct GallStones
Keywords: duodenal-biliary reflux
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recurrent group: Patients with history of recurrent common bile duct stone after successfully ERCP stone remove.
  Interventions: Other: standard barium meal examination
- Control group: Patients without history of recurrent common bile duct stone after successfully ERCP stone remove.
  Interventions: Other: standard barium meal examination

INTERVENTIONS:
Other: standard barium meal examination — All eligible patients received standard barium meal examination, MRCP and enhanced abdominal CT.

SUMMARY:
ERCP is the primary choice for removal of common bile duct stone (CBDS) currently. However, 4-24% patients underwent recurrence after successful clearance of CBDS. Stone re-formation due to chronic inflammation of biliary duct is generally considered an important cause of CBDS recurrence, which is associated with duodenal-biliary reflux (DBR) after sphincterotomy. Although it was believed that DBR was the important cause of CBDS recurrence, the direct evidence was still lacking. Here we conducted a case control study to investigate the DBR rate in patients with recurrent CBDS after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with common bile duct stone underwent successful stone removal by ERCP in Xijing Hospital of Digestive Diseases.

Exclusion Criteria:

* Gallbladder stones or hepatolithiasis;
* Stenosis of biliary duct;
* Incomplete common bile duct stone removal by ERCP;
* Common bile duct stent;
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of recurrent common bile duct stone (recurrent group) and non-recurrent common bile duct stone (control group) in Xijing Hospital of Digestive Diseases were invited to participate the study. All the patients underwent successful stone removal by ERCP previously. Patients in the control group were matched with the recurrence group by age and gender at 1:1 ratio.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Duodenal-biliary reflux rate | up to 6 months
  The proportion of patients with barium reflux into bile duct during the standard barium meal examination.

SECONDARY OUTCOMES:
Distal common bile duct angle | up to 6 months
  MRCP revealed the first angulation from the ampullary orifice along the course of the common bile duct stone.
Maximal CBD diameter | up to 6 months
  Maximal CBD diameter was determined by MRCP.
Peripapillary diverticulum | up to 6 months
  Peripapillary diverticulum was defined endoscopically as the presence of a diverticulum within a 2-cm radius from the papilla and was divided into 2 types in terms of the relation between the papilla and diverticulum: type A, papilla located on the inner rim of the diverticulum or papilla located deep within the diverticulum; and type B, papilla located outside the diverticulum.
Pneumobilia | up to 6 months
  Pneumobilia were determined by CT

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Keizman D, Ish Shalom M, Konikoff FM. Recurrent symptomatic common bile duct stones after endoscopic stone extraction in elderly patients. Gastrointest Endosc. 2006 Jul;64(1):60-5. doi: 10.1016/j.gie.2006.01.022. PMID 16813804
- [Background] Cheon YK, Lehman GA. Identification of risk factors for stone recurrence after endoscopic treatment of bile duct stones. Eur J Gastroenterol Hepatol. 2006 May;18(5):461-4. doi: 10.1097/00042737-200605000-00001. PMID 16607138
- [Background] Ishiguro J. Biliary bacteria as an indicator of the risk of recurrence of choledocholithiasis after endoscopic sphincterotomy. Diagn Ther Endosc. 1998;5(1):9-17. doi: 10.1155/DTE.5.9. PMID 18493475
- [Background] Kim DI, Kim MH, Lee SK, Seo DW, Choi WB, Lee SS, Park HJ, Joo YH, Yoo KS, Kim HJ, Min YI. Risk factors for recurrence of primary bile duct stones after endoscopic biliary sphincterotomy. Gastrointest Endosc. 2001 Jul;54(1):42-8. doi: 10.1067/mge.2001.115335. PMID 11427840
- [Background] Misra SP, Dwivedi M. Reflux of duodenal contents and cholangitis in patients undergoing self-expanding metal stent placement. Gastrointest Endosc. 2009 Aug;70(2):317-21. doi: 10.1016/j.gie.2008.12.054. Epub 2009 Jun 21. PMID 19539920
- [Background] Ando T, Tsuyuguchi T, Okugawa T, Saito M, Ishihara T, Yamaguchi T, Saisho H. Risk factors for recurrent bile duct stones after endoscopic papillotomy. Gut. 2003 Jan;52(1):116-21. doi: 10.1136/gut.52.1.116. PMID 12477771
- [Derived] Zhang R, Luo H, Pan Y, Zhao L, Dong J, Liu Z, Wang X, Tao Q, Lu G, Guo X. Rate of duodenal-biliary reflux increases in patients with recurrent common bile duct stones: evidence from barium meal examination. Gastrointest Endosc. 2015 Oct;82(4):660-5. doi: 10.1016/j.gie.2015.03.1908. Epub 2015 May 5. PMID 25952091